CLINICAL TRIAL: NCT05242835
Title: Management of Sleeve Gastrectomy Failure Using Single-anastomosis Metabolic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Laurent Biertho, Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Second stage SADI
Record Dates: First submitted 2022-01-25; First posted 2022-02-16 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Obesity, Morbid
Keywords: Bariatric surgery
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- biliopancreatic diversion with duodenal switch (Active Comparator): Patient randomized for a the standard duodenal switch as second stage surgery after a sleeve gastrectomy (100cm common channel and 150cm alimentary limb)
  Interventions: Procedure: Standard duodenal switch
- Single-anastomosis duodeno-ileal anastomosis (Experimental): Patient randomized for a single-anastomosis duodeno-ileal anastomosis as second stage surgery after a sleeve gastrectomy (250cm common channel)
  Interventions: Procedure: Single-anastomosis duodenal switch

INTERVENTIONS:
Procedure: Standard duodenal switch — Standard duodenal switch as second stage surgery after a sleeve gastrectomy (100cm common channel and 150cm alimentary limb)
  Other Names: BPD-DS
  Arms: biliopancreatic diversion with duodenal switch
Procedure: Single-anastomosis duodenal switch — Single-anastomosis duodeno-ileal anastomosis as second stage surgery after a sleeve gastrectomy (250cm common channel)
  Other Names: SADI
  Arms: Single-anastomosis duodeno-ileal anastomosis

SUMMARY:
Sleeve gastrectomy (SG) has become the most commonly performed weight loss surgery, accounting for 60% of all bariatric operations worldwide. While technically easier with less side-effects and nutritional risks than other operations, SG is also associated with a higher risk of failure (20 to 40%). In such case, the most effective option consists in adding an intestinal bypass called the Biliopancreatic Diversion with Duodenal Switch (BPD-DS). This surgery is, however, technically challenging and yields a significant risk of complications, nutritional deficiencies or gastro-intestinal side-effects. Recently, a simplified version of the Standard DS, called Single-Anastomosis Duodenoileal Switch (SADI-S) was endorsed by surgical societies as one of the approved bariatric procedures. There is currently no prospective or randomized data to support the effectiveness of this new procedure, especially as a revisional approach. The Overall Objective of this randomized controlled trial project is to establish the clinical benefits of the SADI-S as a revisional surgery after SG, while also considering critical issues related to sex and gender. The investigator Overall Hypothesis is that the SADI-S represents a relevant revisional option for weight loss and metabolic recovery in women and men suffering from severe obesity who had a previous SG. The investigator propose to address the following research question.

Research Question: What are the clinical effects of SADI-S compared to standard DS when used as a revisional procedure after SG, in patients with obesity? Participants who need revisional surgery after SG will be enrolled in a prospective, randomized, double-blind (patient-evaluator), non-inferiority trial comparing SADI-S vs DS. The primary outcome will be 12-month excess weight loss. Secondary outcomes will be perioperative complications, risk of malnutrition, quality of life and gastrointestinal side effects. The investigator hypothesize that SADI-S offers similar weight loss compared to standard DS, but a lower risk of complications and nutritional deficiencies.

With the increase in the number of bariatric operations performed worldwide and the recent endorsement of the SADI-S as a regular procedure, reliable clinical data are urgently needed. The present proposal will directly address this knowledge gap.

ELIGIBILITY:
Inclusion Criteria:

* had sleeve gastrectomy a minimum of 18 months before
* still meet the NIH criteria for bariatric surgery (BMI≥35kg/m2 with major comorbidities or BMI≥40kg/m2) or patients with EWL<50% or significant weight regain (≥20%EWL)

Exclusion Criteria:

* general contra-indication for bariatric surgery
* BMI<35kg/m2
* pregnancy
* cirrhosis
* abnormal bowel habits including irritable bowel syndrome and inflammatory bowel disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Excess weight loss | 12 month
  Percentage of excess weight loss mobilized in response to surgery

SECONDARY OUTCOMES:
Peroperative complications | from baseline up to 60 months
  Complications graded with Clavien classification
Risk of malnutrition | from baseline to 60 months
  Risk of malnutrition assessed through measurement of its risk being mild (albumin<35g\L), moderate (albumin<30g/L) or severe (albumin<25g/L)
Change in quality of life (SF-36) | from baseline to 60 months
  36-item short form survey evaluating quality of life on a scale form 0 to 100
Change in quality of life (BAROS) | from baseline to 60 months
  Bariatric Analyses and Reporting Outcomes System score form -7 to 9
Change in quality of life (QLaval) | from baseline to 60 months
  Laval questionnaire evaluating quality of life on 6 aspects on a scale from 0 to 7
Gastro-intestinal side effects | from baseline to 60 months
  Evaluation of gastro-intestinal side effects with the Gastro-Intestinal Quality of Life Index from 0 to 144
Change in nutritional status (calcium) | from baseline to 60 months
  Change in nutritional status based on blood analysis of calcium (mmol/L)
Change in nutritional status (ferritin) | from baseline to 60 months
  Change in nutritional status based on blood analysis of ferritin (ug/L)
Change in nutritional status (TIBC) | from baseline to 60 months
  Change in nutritional status based on blood analysis of TIBC (umol/L)
Change in nutritional status (iron) | from baseline to 60 months
  Change in nutritional status based on blood analysis of iron (umol/L)
Change in nutritional status (prealbumin) | from baseline to 60 months
  Change in nutritional status based on blood analysis of prealbumin (g/L)
Change in nutritional status (transferrin) | from baseline to 60 months
  Change in nutritional status based on blood analysis transferrin (g/L)
Change in nutritional status (vitamin A) | from baseline to 60 months
  Change in nutritional status based on blood analysis of vitamin A (umol/L)
Change in nutritional status (vitamin D3) | from baseline to 60 months
  Change in nutritional status based on blood analysis of vitamin D3 (nmol/L)
Change in nutritional status (parathormone) | from baseline to 60 months
  Change in nutritional status based on blood analysis parathormone (ng/L)
Change in food intake | from baseline to 60 months
  Evaluation of the change in food intake using a web-based food frequency questionnaire (kcal/day)
Change in eating behavior | from baseline to 60 months
  Change of eating behavior using the Three-Factor Eating Questionnaire evaluating cognitive restraint of eating on a scale from 0 to 20, disinhibition on a scale from 0 to 16 and hunger on a scale from 0 to 15
Change in food addiction | from baseline to 60 months
  Change of eating behavior using the Yale Food Addiction Scale that includes a "symptom count" scale from 0 to 7 reflecting the number of addiction-like criteria endorsed and a dichotomous evaluation that indicates whether a threshold of three or more "symptoms" plus clinically significant impairment or distress has been met
Change in binge eating behavior | from baseline to 60 months
  Change of eating behavior using the Binge Eating scale from 0 to 46
Evolution of obesity related diseases | from baseline to 60 months
  Remission rate for comorbidities, including T2D, hypertension, dyslipidemia, sleep apnea according to the ASMBS definition of outcomes reporting

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Biertho, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec, Canada